CLINICAL TRIAL: NCT02578836
Title: Transoral Gastric Volume Reduction as an Intervention for Weight Management
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was withdrawn due to PI decision
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Roberto Fogel, Associate professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20150200
Record Dates: First submitted 2015-10-15; First posted 2015-10-19 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-05

CONDITIONS: Obesity; Overweight; Weight Loss
Keywords: Weight Loss; Overweight; Endoscopic treatment for obesity
MeSH Terms: conditions — Obesity; Overweight; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fogel Gastroplasty (Experimental): The subject will be placed under general anesthesia. The procedure will last approximately 1-2 hours. CO2 will be used rather than air for the insufflation that is required during the procedure to minimize abdominal distention. The physician will place an interrupted suture pattern in a manner which partitions the greater curvature of the stomach from the Angle of His to the level of the incisura, creating a tube-like passage for gastric volume reduction. Afterwards, the remaining gastric volume will be reduced using a circumferential running stitch.The device that will be used to place the stitches is the OverStitch system FDA approved for tissue apposition
  Interventions: Procedure: Fogel Gastroplasty

INTERVENTIONS:
Procedure: Fogel Gastroplasty — The subject will be placed under general anesthesia. The procedure will last approximately 1-2 hours. CO2 will be used rather than air for the insufflation that is required during the procedure to minimize abdominal distention. The physician will place an interrupted suture pattern in a manner which partitions the greater curvature of the stomach from the Angle of His to the level of the incisura, creating a tube-like passage for gastric volume reduction. Afterwards, the remaining gastric volume will be reduced using a circumferential running stitch.The device that will be used to place the stitches is the OverStitch system FDA approved for tissue apposition
  Other Names: Endoscopic Vertical Gastroplasty

SUMMARY:
This study assesses weight loss from the Endoscopic Vertical Gastroplasty or Fogel Gastroplasty (FG). The purpose of the study is to:

* Document that weight loss occurs (12 months)
* Determine if it alters general wellbeing (emotionally and physically)

DETAILED DESCRIPTION:
This will be a prospective study evaluating the percentage of weight loss in patients that have undergo the Endoscopic Vertical Gastroplasty or Fogel Gastroplasty (FG). Fogel's Gastroplasty is a procedure where The subject will be placed under general anesthesia in accordance with the Institution's standard practice. The procedure will last approximately 1-2 hours. Following induction of anesthesia, the overtube will be placed, a gastroscope will be inserted to examine esophageal and gastric anatomy and re-confirm there are no anatomical contraindications to the procedure. The gastroscope will also be used to record images of the stomach prior to insertion of the OverStitch. Once the examination is complete the gastroscope will be removed. The OverStitch system will then be inserted orally to the per-operative site. CO2 will be used rather than air for the insufflation that is required during the procedure to minimize abdominal distention. The physician will place an interrupted suture pattern in a manner which partitions the greater curvature of the stomach from the Angle of His to the level of the incisura, creating a tube-like passage for gastric volume reduction. Afterwards, the remaining gastric volume will be reduced using a circumferential running stitch. Once complete, the OverStitch system will be removed and a standard gastroscope will be inserted to record post procedure endoscopic images.

Anthropometric measurements as Weight, Height, BMI and Waist Circumference will be collected at Baseline, 3, 6 and 12 months after procedure

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 yrs. of age and ≤ 60 yrs. of age
2. Subject has a BMI between 28 and 34.9
3. Subject is willing to complete all follow-up visits after procedure ( 3, 6 and 12 months)

Exclusion Criteria:

1. Patients that are not willing to participate in the study
2. Patients with history of Gastrointestinal tumors, Gastric Cancer, previous bariatric, gastric or esophageal surgery; intestinal obstruction; portal gastropathy, esophageal or gastric varices, or gastroparesis,
3. Subject has significant esophageal disease including Zenker's diverticulum, grade 3-4 reflux esophagitis, stricture, Barrett's esophagus, esophageal cancer, esophageal diverticulum, dysphagia, achalasia, or symptoms of dysmotility or Hiatal Hernia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2018-03 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Weight Loss | 12 months

SECONDARY OUTCOMES:
Emotional Wellbeing | 12 months
  Measured by self administration of quality of life questionnaire SF-36
Change in blood pressure | baseline to 12 months
Change in cholesterol level | baseline to 12 months
Change in glucose levels | baseline to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Fogel, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Clinical Research Building, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided